CLINICAL TRIAL: NCT00032006
Title: A Trial Of Neoadjuvant Androgen Supression And Dose Escalation Transperineal Ultrasound-Guided Brachytherapy For Locally Recurrent Prostate Adenocarcinoma Following External Beam Radiotherapy
Brief Title: Hormone Therapy Followed By Internal Radiation Therapy in Treating Patients With Locally Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0052; CDR0000069248 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- brachytherapy + radiation (Experimental): Within 4 weeks after completion of androgen suppression, patients are sequentially enrolled to 2 different cohorts of brachytherapy.
  Cohort 1: Patients undergo initial-dose transperineal interstitial permanent prostate brachytherapy with iodine I 125 or palladium Pd 103.
  Cohort 2: After a minimum of 1-year follow-up for all patients in cohort 1, if tolerance is acceptable, additional patients undergo higher-dose transperineal interstitial permanent prostate brachytherapy with iodine I 125 or palladium Pd 103.
  Quality of life is assessed at baseline, within 2 weeks prior to brachytherapy, every 3 months for 1 year, and then every 6 months for 2 years.
  Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.
  Interventions: Radiation: brachytherapy; Radiation: radiation therapy

INTERVENTIONS:
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as goserelin, leuprolide, flutamide, or bicalutamide may stop the adrenal glands from producing androgens. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Combining hormone therapy with internal radiation may be effective in treating locally recurrent prostate cancer.

PURPOSE: Phase II trial to study the effectiveness of hormone therapy followed by internal radiation in treating patients who have locally recurrent prostate cancer following external-beam radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the nature, intensity, and time course of health-related quality of life changes in patients with locally recurrent prostate adenocarcinoma treated with androgen suppression and transperineal ultrasound-guided brachytherapy after external beam radiotherapy.
* Determine the morbidity of patients treated with this regimen.
* Determine the overall survival, disease-free survival, and disease-specific survival of patients treated with this regimen.
* Determine the clinical patterns of tumor recurrence (i.e., time to local tumor progression or distant failure) and time to biochemical failure of patients treated with this regimen.
* Determine the post-brachytherapy dosimetric coverage of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive androgen suppression comprising goserelin subcutaneously (as either 4 one-month depot injections or 1 one-month depot injection and 1 three-month depot injection) OR leuprolide intramuscularly (as 4 one-month depot injections or 1 one-month depot injection and 1 three-month depot injection or 1 four-month depot injection) AND oral flutamide 3 times daily for 112 days OR oral bicalutamide once daily for 112 days.

Within 4 weeks after completion of androgen suppression, patients are sequentially enrolled to 2 different cohorts of brachytherapy.

* Cohort 1: Patients undergo initial-dose transperineal interstitial permanent prostate brachytherapy with iodine I 125 or palladium Pd 103.
* Cohort 2: After a minimum of 1-year follow-up for all patients in cohort 1, if tolerance is acceptable, additional patients undergo higher-dose transperineal interstitial permanent prostate brachytherapy with iodine I 125 or palladium Pd 103.

Quality of life is assessed at baseline, within 2 weeks prior to brachytherapy, every 3 months for 1 year, and then every 6 months for 2 years.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 83-166 patients (83 per cohort) will be accrued for this study within 1.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally recurrent or persistent prostate adenocarcinoma

  * Locally recurrent disease
  * Prostate-specific antigen (PSA) no greater than 10 ng/mL
  * N0 and M0 (at time of initial diagnosis and at time of local recurrence)

    * Lymph nodes must be negative or will be negative after nodal sampling or dissection
* More than 18 months after completion of prior external beam radiotherapy
* Must have had 1 of the following disease characteristics prior to external beam radiotherapy:

  * T1-2a, Gleason score 2-6, and PSA no greater than 15 ng/mL
  * T1-2a, Gleason score 7, and PSA no greater than 4 ng/mL
  * T2b, Gleason score 2-6, and PSA no greater than 6 ng/mL
* Must have American Urological Association Symptom Index score no greater than 15
* Transrectal ultrasound-determined prostate planimetry volume no greater than 60 mL
* No pubic arch interference of more than 1/3 the prostatic volume determined by transrectal ultrasound or pelvic CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1 OR
* ECOG 0-1

Life expectancy:

* At least 5 years

Other:

* No persistent late intestinal or bladder toxicity grade 2 or greater
* No other major medical or psychiatric illness that would preclude study
* No metallic hip prosthesis
* No other malignancy within the past 5 years except localized basal cell or squamous cell skin cancer
* No other concurrent illness that would limit life expectancy
* Suitable for spinal or general anesthesia
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* No prior chemotherapy for prostate cancer

Endocrine therapy:

* At least 12 months since prior androgen suppression except goserelin or leuprolide with flutamide or bicalutamide begun within the past 30 days

Radiotherapy:

* See Disease Characteristics
* No prior external beam radiotherapy doses exceeding 71 Gy to the prostate
* No prior radionuclide prostate brachytherapy

Surgery:

* No prior transurethral prostate resection
* No prior prostatectomy or prostatic cryosurgery
* No prior bilateral orchiectomy

Other:

* No concurrent participation in another medical research study for prostate cancer treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-02; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
quality of life | Up to 10 years

SECONDARY OUTCOMES:
Morbidity | Up to 10 years
Disease free survival | Up to 10 years
Disease specific survival | Up to 10 years
tumor recurrence | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Pisansky, MD, Study Chair — Mayo Clinic
Locations (8):
- United States (8):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin